CLINICAL TRIAL: NCT02389335
Title: Roles of Interferon Gamma, Interleukin-2 and Tumor Necrotizan Factor Alpha in the Pathogenesis of Type 1 Diabetes
Brief Title: Roles of T Helper 1 Cytokines in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gonca Incemehmet Tamer, Assoc prof, Istanbul Medeniyet University
Other Study IDs: MUGEAH-2; Interleukins in type 1diabetes (Registry Identifier: Interleukins)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Type 1 Diabetes
Keywords: type 1diabetes; IFN γ; IL-2; TNF α
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1a: Patients with type 1 diabetes who have undetectable c-peptide ( ≤0.1 ng/mL) levels after mixed meal tolarance test: group 1a
- Group 1b: Patients with type 1 diabetes who have c-peptide levels between 0.1-0.8 ng/mL after mixed meal tolerance test: group 1b
- Group 1c: Patients with type 1 diabetes who have c-peptide levels ≥0.8ng/mL after mixed meal tolerance test: group 1c
- Control: Healthy subjects

SUMMARY:
The mechanism of β cell destruction in Type 1 diabetes is not exactly known, Our hyphotesis is that interferon gamma, interleukin-2 and tumor necrotizan factor alpha have impotant roles in β cell destruction.

DETAILED DESCRIPTION:
T helper (h)1 cells are known to have important roles in the destruction or/and dedifferentiation of β-cells in type 1 diabetes (T1D). Significant increase in IFN-γ-producing Th1 cells in the pancreas and in the serum levels were determined in type 1 diabetic patients at diabetes oneset. This data indicated that this proinflammatory mediator serve as a biomarker of advanced autoimmunity. We aimed to investigate the relationship between Th1 cytokines (IFN-γ, IL-2 and TNF-α) and T1D and the effect of those cytokines on β-cell function.

ELIGIBILITY:
Inclusion Criteria:

* Patients giving consent to participate the study
* Patients with type 1 diabetes according to WHO definiton

Exclusion Criteria:

* Acute and chronic inflammatory diseases,
* significant concomitant diseases which may interfere with glucose metabolism
* cancers,
* hemoglobinopathies,
* recently received antibiotics,
* drugs influencing β-cell function and
* insulin sensitivity or anti-inflammatory drugs
* recent history of trauma

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study included 98 T1DPs and 30 healthy subjects (CG). All subjects
  were matched on age and gender. β-cell function of 98 T1DPS was assesseed by measuring C-Peptide levels
  after mixed-meal tolarence test (MMTT)s. T1DPs were divided into 3
  groups according to the C-Peptide levels after MMTTs and the groups
  were as follows: patients with undetectable ≤0.1 ng/mL(group 1a, n=30)
  C-Peptide levels; minimal 0.1-0.8 ng/mL(group1b, n=30); and sustained
  ≥0.8ng/mL(group1c, n=38) C-peptide levels which increased at the 90th
  minute after the meal ≥150% of fasting C-peptide level.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Roles of interferon gamma, interleukin-2, tumor necrotizan factor alpha in the pathogenesis of type 1 diabetes | 3 day

CONTACTS AND LOCATIONS:
Locations (1):
- Medeniyet University Goztepe Training and Research Hospital, Istanbul, Turkey (Türkiye)